CLINICAL TRIAL: NCT04294459
Title: A Phase 1b/2 Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of Isatuximab (SAR650984) in Patients Awaiting Kidney Transplantation
Brief Title: Safety, Pharmacokinetics, and Preliminary Efficacy of Isatuximab in Patients Awaiting Kidney Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to non-safety reasons
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED16414; 2019-004154-28 (EudraCT Number); U1111-1238-9716 (Other: UTN)
Record Dates: First submitted 2020-02-19; First posted 2020-03-04 (Actual); Results first posted 2023-05-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Immune System Disorder
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Immune System Diseases | interventions — isatuximab; Acetaminophen; Ranitidine; Diphenhydramine; Methylprednisolone; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Participants with cPRA >=99.90% (Experimental): Participants with calculated panel reactive antibodies (cPRA) >=99.90% (indicating active candidates on kidney transplant waitlist) received isatuximab 10 milligrams per kilogram (mg/kg), intravenous (IV) infusion, once weekly (QW) for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1) and then every 2 weeks (Q2W) for subsequent treatment cycles (each cycle of 28 days) until unacceptable adverse events (AEs) or participant's decision to stop the treatment (maximum treatment duration: 13 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Acetaminophen (paracetamol) or equivalent; Drug: Ranitidine or equivalent; Drug: Diphenhydramine or equivalent; Drug: Methylprednisolone or equivalent; Drug: Montelukast or equivalent
- Cohort B: Participants with cPRA 80.00% to 99.89% (Experimental): Participants with cPRA between 80.00% to 99.89% (indicating active candidates on kidney transplant waitlist with no living donor cleared for donation) received isatuximab 10 mg/kg, IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1) and then Q2W for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs or participant's decision to stop the treatment (maximum treatment duration: 13 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Acetaminophen (paracetamol) or equivalent; Drug: Ranitidine or equivalent; Drug: Diphenhydramine or equivalent; Drug: Methylprednisolone or equivalent; Drug: Montelukast or equivalent

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: Solution for infusion
  Route of administration: Intravenous
  Other Names: Sarclisa
Drug: Acetaminophen (paracetamol) or equivalent — Pharmaceutical form: Tablets
  Route of administration: Oral
Drug: Ranitidine or equivalent — Pharmaceutical form: Solution
  Route of administration: Intravenous
Drug: Diphenhydramine or equivalent — Pharmaceutical form: Solution
  Route of administration: Intravenous
Drug: Methylprednisolone or equivalent — Pharmaceutical form: Solution
  Route of administration: Intravenous
Drug: Montelukast or equivalent — Pharmaceutical form: Tablets
  Route of administration: Oral

SUMMARY:
Primary Objectives:

* Phase 1: To characterize the safety and tolerability of isatuximab in kidney transplant candidates.
* Phase 2: To evaluate the efficacy of isatuximab in desensitization of participants awaiting kidney transplantation.

Secondary Objectives:

* Phase 2: To characterize the safety profile of isatuximab in kidney transplant candidates.
* To characterize the pharmacokinetic (PK) profile of isatuximab in kidney transplant candidates.
* To evaluate the immunogenicity of isatuximab.
* To assess the overall efficacy of isatuximab in desensitization of participants awaiting kidney transplantation.

DETAILED DESCRIPTION:
The study had a screening period of up to 28 days, a treatment period of up to 12 weeks, a site visit FUP of up to 26 weeks, and an extended follow-up (FUP) until study cut-off.

The study duration involved site visit per participant (i.e., screening, treatment, site visit FUP was approximately 42 weeks.

The study duration included extended FUP per participant was approximately 97.7 weeks (depending on when the participant was enrolled).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of chronic kidney disease (CKD) and active candidate on the kidney donor waitlist at the time of screening.
* Body mass index (BMI) </=40 kg/m^2.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

For Participants in Cohort A: active candidates on the kidney waitlist with living donor.

For Participants in Cohort B: active candidates on the kidney waitlist with no living donor cleared for donation.

Exclusion criteria:

* Significant cardiac dysfunction.
* Known active, recurrent, or chronic infection.
* Active lupus or uncontrolled diabetes.
* Prior treatment with rituximab within 6 months from SAR650984 administration.
* Inadequate organ and bone marrow function at screening.
* Pregnant or breastfeeding women or women who intend to become pregnant during participation in the study.
* Known intolerance or hypersensitivity to any component of SAR650984 or pre-medications.
* Participants who were not suitable for participation as judged by the Investigator.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (4):
  - Investigational Site Number :8400003, San Francisco, California
  - Investigational Site Number :8400001, Rochester, Minnesota
  - Investigational Site Number :8400002, New York, New York
  - Investigational Site Number :8400004, Houston, Texas
- Spain (2):
  - Investigational Site Number :7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240001, L'Hospitalet de Llobregat, Catalunya [Cataluña]

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Mannon RB, Vincenti FG. Poised for Innovation: Considerations for End Points for New Drug Development in Kidney Transplantation. J Am Soc Nephrol. 2024 Nov 1;35(11):1603-1606. doi: 10.1681/ASN.0000000000000475. Epub 2024 Aug 5. No abstract available. PMID 39102302
- [Derived] Vincenti F, Bestard O, Brar A, Cruzado JM, Seron D, Gaber AO, Ali N, Tambur AR, Lee H, Abbadessa G, Paul JA, Dudek M, Siegel RJ, Torija A, Semiond D, Lepine L, Ternes N, Montgomery RA, Stegall M. Isatuximab Monotherapy for Desensitization in Highly Sensitized Patients Awaiting Kidney Transplant. J Am Soc Nephrol. 2024 Mar 1;35(3):347-360. doi: 10.1681/ASN.0000000000000287. Epub 2023 Dec 26. PMID 38147137
- See also: TED16414 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25360&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 6 active sites in 2 countries. A total of 23 participants were enrolled between 18 Jun 2020 and 02 Nov 2021 and received isatuximab monotherapy.
Pre-assignment Details: Study was planned to be conducted in 2 parts: Phase 1 (safety run-in) and Phase 2 (efficacy). Sponsor decided to terminate the study for non-safety reasons on 02 May 2022. Based on available clinical data at time of interim analysis, it was determined that enrollment of remaining participants was unlikely to have any significant impact on study results and hence trial was stopped. Participant flow, baseline, outcome measures and safety data were presented for combined Phase 1 and 2 population.
Period: Overall Study
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Cohort A: Participants With cPRA >=99.90%: Participants with cPRA >=99.90%; (indicating active candidates on kidney transplant waitlist) received isatuximab 10 mg/kg, IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1) and then Q2W for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs or participant's decision to stop the treatment (maximum treatment duration: 13 weeks).
- Total: Total of all reporting groups
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89% | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.9) | 48.2 (12.3) | 49.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 4 | 9 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious adverse events (SAEs) were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (defined as the time from the first dose of study drug until study cut-off date).
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on all treated population which included all participants who received at least one dose of isatuximab. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Participants With cPRA >=99.90%: Participants with cPRA >=99.90% (indicating active candidates on kidney transplant waitlist) received isatuximab 10 mg/kg, IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1) and then Q2W for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs or participant's decision to stop the treatment (maximum treatment duration: 13 weeks).
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  TEAEs | 3 | 4
  TESAEs | 0 | 0

2. Primary Outcome: Number of Participants With Hematological Abnormalities
Description: Abnormal hematological parameters assessed were anemia, platelet count decreased, neutrophil count decreased, lymphocyte count decreased and monocytes. The hematological abnormality grades were based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs. Monocytes were assessed as per potentially clinically significant abnormality (PCSA) criteria defined as: greater than (>) 0.7*10^9/L.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on all treated population. Here, "number analyzed" = participants with available data for each specified category. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  Anemia: Grade 1 | 6 | 8
  Anemia: Grade 2 | 3 | 2
  Anemia: Grade 3 | 0 | 0
  Anemia: Grade 4 | 0 | 0
  Platelet count decreased: Grade 1 | 2 | 6
  Platelet count decreased: Grade 2 | 0 | 0
  Platelet count decreased: Grade 3 | 0 | 0
  Platelet count decreased: Grade 4 | 0 | 0
  Neutrophil count decreased: Grade 1: number analyzed (Participants) | 9 | 7
  Neutrophil count decreased: Grade 1 | 0 | 0
  Neutrophil count decreased: Grade 2: number analyzed (Participants) | 9 | 7
  Neutrophil count decreased: Grade 2 | 0 | 0
  Neutrophil count decreased: Grade 3: number analyzed (Participants) | 9 | 7
  Neutrophil count decreased: Grade 3 | 0 | 0
  Neutrophil count decreased: Grade 4: number analyzed (Participants) | 9 | 7
  Neutrophil count decreased: Grade 4 | 0 | 0
  Lymphocyte count decreased: Grade 1: number analyzed (Participants) | 9 | 7
  Lymphocyte count decreased: Grade 1 | 4 | 2
  Lymphocyte count decreased: Grade 2: number analyzed (Participants) | 9 | 7
  Lymphocyte count decreased: Grade 2 | 1 | 1
  Lymphocyte count decreased: Grade 3: number analyzed (Participants) | 9 | 7
  Lymphocyte count decreased: Grade 3 | 1 | 0
  Lymphocyte count decreased: Grade 4: number analyzed (Participants) | 9 | 7
  Lymphocyte count decreased: Grade 4 | 0 | 0
  Monocytes (PCSA) > 0.7*10^9/L: number analyzed (Participants) | 9 | 7
  Monocytes (PCSA) > 0.7*10^9/L | 3 | 3

3. Primary Outcome: Number of Participants With Renal Function Abnormalities
Description: Abnormal renal parameters assessed were creatinine increased and estimated Glomerular Filtration Rate (eGFR). The renal function abnormality grades were based on NCI-CTCAE, Version 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs. eGFR was assessed as per PCSA criteria: 60 (less than equal to) <= to less than (<) 90 milliliter/minute/1.73 meter square (mL/min/1.73m^2) (Mild), 30<= to <60 mL/min/1.73m^2 (Moderate), 15<=to <30 mL/min/1.73m^2 (Severe), <15 mL/min/1.73m^2 (End Stage Renal Disease).
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on all treated population. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  Creatinine increased: Grade 1 | 0 | 0
  Creatinine increased: Grade 2 | 0 | 0
  Creatinine increased: Grade 3 | 1 | 3
  Creatinine increased: Grade 4 | 11 | 8
  eGFR: 60<= - <90 mL/min/1.73m^2 | 0 | 0
  eGFR: 30<= - <60 mL/min/1.73m^2 | 0 | 0
  eGFR: 15<= - <30 mL/min/1.73m^2 | 0 | 0
  eGFR: <15 mL/min/1.73m^2 | 12 | 11

4. Primary Outcome: Number of Participants With Abnormal Electrolytes Parameters
Description: Abnormal electrolyte parameters assessed were hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypercalcemia, hypocalcemia, blood bicarbonate decreased, hypermagnesemia, hypomagnesemia and chloride. The abnormal grades were based on NCI-CTCAE, Version 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs. Chloride was estimated as per PCSA criteria: <80 millimoles per liter (mmol/L) and >115 mmol/L.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on all treated population. Here, 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field signifies that none of the participants were available for assessment of the specified parameter. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  Hypernatremia: Grade 1 | 0 | 0
  Hypernatremia: Grade 2 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0
  Hyponatremia: Grade 1 | 4 | 1
  Hyponatremia: Grade 2 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 0
  Hyponatremia: Grade 4 | 0 | 0
  Hyperkalemia: Grade 1 | 2 | 6
  Hyperkalemia: Grade 2 | 3 | 1
  Hyperkalemia: Grade 3 | 1 | 2
  Hyperkalemia: Grade 4 | 0 | 0
  Hypokalemia: Grade 1 | 0 | 0
  Hypokalemia: Grade 2 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 0
  Hypokalemia: Grade 4 | 1 | 0
  Hypercalcemia: Grade 1 | 0 | 1
  Hypercalcemia: Grade 2 | 1 | 0
  Hypercalcemia: Grade 3 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0
  Hypocalcemia: Grade 1 | 6 | 5
  Hypocalcemia: Grade 2 | 0 | 2
  Hypocalcemia: Grade 3 | 0 | 0
  Hypocalcemia: Grade 4 | 0 | 0
  Blood bicarbonate decreased: Grade 1: number analyzed (Participants) | 0 | 0
  Blood bicarbonate decreased: Grade 2: number analyzed (Participants) | 0 | 0
  Blood bicarbonate decreased: Grade 3: number analyzed (Participants) | 0 | 0
  Blood bicarbonate decreased: Grade 4: number analyzed (Participants) | 0 | 0
  Hypermagnesemia: Grade 1 | 2 | 0
  Hypermagnesemia: Grade 2 | 0 | 0
  Hypermagnesemia: Grade 3 | 0 | 0
  Hypermagnesemia: Grade 4 | 0 | 0
  Hypomagnesemia: Grade 1 | 3 | 3
  Hypomagnesemia: Grade 2 | 0 | 0
  Hypomagnesemia: Grade 3 | 0 | 0
  Hypomagnesemia: Grade 4 | 0 | 0
  Chloride (PCSA): <80 mmol/L | 0 | 0
  Chloride (PCSA): >115 mmol/L | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Metabolism Parameters
Description: Abnormal metabolism parameters assessed were hypoglycemia, hypoalbuminemia and glycated Hemoglobin (HbA1c). The abnormal grades were based on NCI-CTCAE, Version 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs. HbA1c was estimated as per PCSA criteria: >8%.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on all treated population. Here, "number analyzed" = participants with available data for each specified category and "0" in the number analyzed field signifies that none of the participants were available for assessment of the specified parameter. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  Hypoglycemia: Grade 1 | 1 | 2
  Hypoglycemia: Grade 2 | 1 | 0
  Hypoglycemia: Grade 3 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0
  Hypoalbuminemia: Grade 1 | 3 | 0
  Hypoalbuminemia: Grade 2 | 2 | 2
  Hypoalbuminemia: Grade 3 | 0 | 0
  Hypoalbuminemia: Grade 4 | 0 | 0
  HbA1c (PCSA): number analyzed (Participants) | 0 | 0

6. Primary Outcome: Number of Participants With Liver Function Abnormalities
Description: Abnormal liver function parameters assessed were Alanine aminotransferase (ALT) increased, Aspartate aminotransferase (AST) increased, Alkaline phosphatase (ALP) increased, and Total bilirubin (TB) increased. The abnormal grades were based on NCI-CTCAE, Version 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  ALT increased: Grade 1 | 1 | 1
  ALT increased: Grade 2 | 0 | 0
  ALT increased: Grade 3 | 0 | 0
  ALT increased: Grade 4 | 0 | 0
  AST increased: Grade 1 | 1 | 0
  AST increased: Grade 2 | 0 | 0
  AST increased: Grade 3 | 0 | 0
  AST increased: Grade 4 | 0 | 0
  ALP increased: Grade 1 | 3 | 2
  ALP increased: Grade 2 | 0 | 0
  ALP increased: Grade 3 | 0 | 0
  ALP increased: Grade 4 | 0 | 0
  TB increased: Grade 1 | 0 | 0
  TB increased: Grade 2 | 0 | 0
  TB increased: Grade 3 | 0 | 0
  TB increased: Grade 4 | 0 | 0

7. Primary Outcome: Percentage of Participants With Response
Description: Response was defined as the percentage of participants meeting at least one of the predefined desensitization efficacy criteria as measured by single antigen bead (SAB) assay as follows: reduction in cPRA resulting in at least 100% increase of likelihood of finding a compatible donor; reduction in antibody titer (>=75% reduction from Baseline) to achieve target cPRA; elimination of >=1 human leukocyte antigen (HLA) antibody (i.e., mean fluorescence intensity [MFI] reduced to <2000) as measured by a SAB assay, for antibodies with Baseline MFI >=3000.
Time Frame: From first dose of study drug until end of follow-up period (maximum duration: up to 39.1 weeks)
Population: Analysis was performed on efficacy evaluable population which included all participants who received at least 1 dose of isatuximab, with an evaluable Baseline and at least 1 evaluable post-baseline efficacy assessment and received >=75% of planned cumulative doses. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
percentage of participants | 83.3 [51.6 to 97.9] | 81.8 [48.2 to 97.7]

8. Secondary Outcome: Pharmacokinetics (PK) Parameters: Concentration Observed at the End of First Intravenous Infusion (Ceoi) of Isatuximab
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion of isatuximab.
Time Frame: At End of infusion on Cycle 1 Day 1
Population: Analysis was performed on pharmacokinetic (PK) population which included all participants who receive at least 1 dose of isatuximab, with at least 1 available concentration result post treatment. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 11 | 11
micrograms per milliliter (mcg/mL) | 290 (128) | 270 (101)

9. Secondary Outcome: PK Parameters: Maximum Concentration Observed (Cmax) After the First Infusion of Isatuximab
Description: Cmax was defined as the maximum concentration observed after the first administration calculated using the noncompartmental analysis after the intravenous infusion of isatuximab.
Time Frame: At Start of infusion (SOI), End of infusion (EOI), EOI+4H (initial protocol) EOI+1H (amended protocol), 72H and 168H on Day 1 of Cycle 1
Population: Analysis was performed on PK population. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 11 | 11
mcg/mL | 295 (128) | 285 (94.0)

10. Secondary Outcome: PK Parameters: Time Taken to Reach Cmax (Tmax) After the First Infusion of Isatuximab
Description: Tmax was defined as the time to reach Cmax, calculated using the non-compartmental analysis after the intravenous infusion of isatuximab.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 11 | 11
hours | 3.67 [2.00 to 6.03] | 3.40 [2.25 to 4.63]

11. Secondary Outcome: PK Parameters: Last Concentration Observed Above the Lower Limit of Quantification (Clast) After the First Infusion of Isatuximab
Description: Clast was defined as the last concentration of isatuximab observed above the lower limit of quantification calculated using non-compartmental analysis after the first infusion of isatuximab.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 11 | 11
mcg/mL | 104 (41.7) | 76.3 (21.3)

12. Secondary Outcome: PK Parameters: Time of Clast (Tlast) After First Infusion of Isatuximab
Description: Tlast was defined as the time of last concentration observed above the lower limit of quantification, calculated using the non-compartmental analysis after the intravenous infusion of isatuximab.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 11 | 11
hours | 166.00 [49.60 to 169.00] | 167.00 [78.80 to 168.00]

13. Secondary Outcome: PK Parameters: Trough Plasma Concentrations (Ctrough) of Isatuximab
Description: Ctrough was the plasma concentration of isatuximab observed just before (pre-dose) treatment administration.
Time Frame: Cycle 2 Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 11 | 10
mcg/mL | 308 (79.4) | 246 (60.6)

14. Secondary Outcome: PK Parameters: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 168 Hours Over the Dosing Interval (AUC0-168 Hours) After First Infusion of Isatuximab
Description: AUC0-168 hours was defined as the area under the plasma concentration versus time curve from time 0 to 168 hours post dose calculated using trapezoidal method after first infusion of isatuximab.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micrograms*hours/milliliter (mcg*h/mL)
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 10 | 10
micrograms*hours/milliliter (mcg*h/mL) | 29400 (7400) | 20000 (5240)

15. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Against Isatuximab
Description: ADA responses were categorized as treatment boosted ADA and treatment-induced ADA. Treatment boosted ADA was defined as pre-existing ADAs with a significant increase in the ADA titer during the study compared to the Baseline titer. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on anti-drug antibodies (ADA) population which included all participants who receive at least 1 dose of isatuximab, with at least 1 available ADA result post-treatment. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  Treatment-induced ADA | 0 | 0
  Treatment boosted ADA | 0 | 0

16. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was defined as time (in weeks) from laboratory sample collection date used in determining a participant to be a responder (defined as participants meeting at least one of the predefined desensitization efficacy criteria: reduction in cPRA resulting in at least 100% increase of likelihood of finding a compatible donor; reduction in antibody titer [>=75% reduction from Baseline] to achieve target cPRA; elimination of >=1 anti-HLA antibody i.e. MFI reduced to <2000 as measured by a SAB assay, for antibodies with Baseline MFI >=3000) up to the laboratory sample collection date when participant was confirmed as no longer meeting any response criterion (i.e., non-responder) or the date of death due to any cause, whichever occurs first. DOR was analyzed using Kaplan-Meier method.
Time Frame: From first dose of study drug until end of follow-up period (maximum duration: up to 39.1 weeks)
Population: Analysis was performed on responder population which included all participants who received at least 1 dose of isatuximab, with an evaluable Baseline and at least 1 evaluable post-baseline efficacy assessment and received >=75% of planned cumulative doses. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 10 | 9
weeks | NA [4.857 to NA] — Due to insufficient number of participants with events, median DOR and upper limit of confidence interval (CI) was not reached. | NA [4.143 to NA] — Due to insufficient number of participants with events, median DOR and upper limit of CI was not reached.

17. Secondary Outcome: Number of Participants Achieving Target cPRA
Description: Target calculated panel reactive antibodies (cPRA) was defined as the reduction of cPRA required to achieve at least 100% increase of likelihood of compatible donor (LCD). Number of participants who achieved target cPRA was assessed using the Organ Procurement and Transplantation Network (OPTN) calculator during the specified timepoint were reported in this outcome measure. Participants who retained their target cPRA values were censored at the date of the last available laboratory assessment achieving their target cPRA.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on efficacy evaluable population. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 7 | 6
Participants | 4 | 2

18. Secondary Outcome: Duration for Achieving Target cPRA
Description: Duration of achieving target cPRA was defined as the time (in weeks) from laboratory sample collection date of achieving target cPRA (defined as the reduction of cPRA required to achieve at least 100% increase of LCD) the first time up to the laboratory sample collection date when no longer achieving target cPRA calculated using OPTN calculator or the date of death due to any cause, whichever occurs first. The duration of achieving target cPRA was assessed using the Kaplan-Meier method.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 4 | 2
weeks | NA [3.429 to NA] — Due to insufficient number of participants with events, median and upper limit of CI was not reached. | 7.29 [NA to NA] — Due to insufficient number of participants with events, upper and lower limit of CI was not reached.

19. Secondary Outcome: Number of Participants With Anti-Human Leukocyte Antigen (HLA)-Antibody Reduction
Description: Number of participants with anti-HLA-antibody (Baseline MFI >=3000) reduced to <2000 as measured using a SAB assay per central laboratory assessment was reported in this outcome measure. Participants were categorized in various categories of number of antibodies which were reduced as: none, 1-5, >5-10, >10-15, and >15. If multiple visits had the same number of total anti-HLA antibody reduction, the last visit data was summarized.
Time Frame: From first dose of study drug until end of follow-up period (maximum duration: up to 39.1 weeks)
Population: Analysis was performed on efficacy evaluable population. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
Participants
  None | 2 | 2
  1-5 antibodies | 4 | 4
  >5-10 antibodies | 4 | 4
  >10-15 antibodies | 1 | 0
  >15 antibodies | 1 | 1

20. Secondary Outcome: Time to First Transplant Offer
Description: Time to first transplant offer was defined as time (in days) from date of first study treatment dose up to date of first kidney transplant offer. Data on transplant status were collected and followed up until study cut-off date.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on efficacy-evaluable population. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 3 | 3
days | 373 [248 to 517] | 156 [117 to 402]

21. Secondary Outcome: Time to Transplant
Description: Time to transplant was defined as time (in days) from date of first study treatment dose up to date of kidney transplant. Data on transplant status were collected and followed up until study cut-off date.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on efficacy evaluable population. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure and included only participants who accepted transplant offer. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 2 | 2
days | 445 [373 to 517] | 259.5 [117 to 402]

22. Secondary Outcome: Number of Kidney Transplant Offers
Description: Number of kidney transplants offers received for each participant was reported in the outcome measure. Data on transplant offers were collected and followed up until study cut-off date.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Analysis was performed on efficacy-evaluable population. Data was planned to be collected and analyzed for the combined Phase 1 and 2 population.
Measure: Number; unit: transplant offers
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
Number analyzed (Participants) | 12 | 11
transplant offers | 3 | 3

23. Secondary Outcome: Time to First Antibody Mediated Rejection (AMR) Episode
Description: Time to first AMR was defined as time from date of first study treatment dose up to date of biopsy with first AMR (defined as the graft rejection due to generation of antibodies against the graft). Transplanted participants without any AMR were censored at the participant's last assessment or contact date collected in the study or at the analysis cut-off date, whichever was earlier.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Data for this outcome measure was not collected and analyzed as no participants experienced a kidney transplant graft loss due to an AMR episode as of study terminated date.
Groups:
- Cohort B: Participants With Calculated Panel Reactive Antibodies (cPRA) 80.00% to 99.89%: Participants with cPRA between 80.00% to 99.89% (indicating active candidates on kidney transplant waitlist with no living donor cleared for donation) received isatuximab 10 mg/kg, IV infusion, QW for 4 weeks (i.e., on Day 1, Day 8, Day 15 and Day 22 of Cycle 1) and then Q2W for subsequent treatment cycles (each cycle of 28 days) until unacceptable AEs or participant's decision to stop the treatment (maximum treatment duration: 13 weeks).
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With Calculated Panel Reactive Antibodies (cPRA) 80.00% to 99.89%
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Percentage of Participants Who Experienced Any Antibody Mediated Rejection (AMR)
Description: Antibody mediated rejection was defined as the graft rejection due to generation of antibodies against the graft. The number of participants with AMR field checked as 'yes' based on the graft rejection biopsy in the electronic case report form was considered.
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Population: Data for this outcome measure was not collected and analyzed as no participants experienced a kidney transplant graft loss due to an AMR episode, as of study terminated date.
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With Calculated Panel Reactive Antibodies (cPRA) 80.00% to 99.89%
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Number of Participants With Graft Survival at 6 Months Post-Transplant
Description: Number of participants with graft survival status as functioning at 6-months post-transplant was reported in this outcome measure.
Time Frame: At 6 Months post-transplant
Population: Analysis was performed on efficacy evaluable population. Here, "overall number of participants analyzed" signifies participants with evaluable data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With Calculated Panel Reactive Antibodies (cPRA) 80.00% to 99.89%
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until study cut-off date (maximum duration: up to 97.7 weeks)
Description: Analysis was performed on all treated population.
Arm/Group | Cohort A: Participants With cPRA >=99.90% | Cohort B: Participants With cPRA 80.00% to 99.89%
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 3/12 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Participants With cPRA >=99.90% (N=12) | Cohort B: Participants With cPRA 80.00% to 99.89% (N=11)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
Sponsor decided to terminate the study for non-safety reasons on 02 May 2022. Based on available clinical data at time of interim analysis, it was determined that enrollment of the remaining participants was unlikely to have any significant impact on the study results and hence the trial was stopped. All 23 participants enrolled in the study were followed-up per protocol until the planned study termination date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04294459/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT04294459/SAP_001.pdf